CLINICAL TRIAL: NCT06465173
Title: Is Self-compassion Associated With Older Adults' Quality of Life After Dementia Diagnosis and Does Perceived Threat Posed by Dementia Mediate This Relationship?
Brief Title: Self-compassion and Quality of Life After Dementia Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Oxford Health NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PID 17089
Record Dates: First submitted 2024-05-24; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Dementia
Keywords: dementia; self-compassion; quality of life
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 'High self-compassion' group: Participants' total mean score on the Self-compassion Scale - Short Form (Raes et al., 2011) will be used as the independent variable. A median split (+/-1 standard error of the median) on the Self-compassion Scale - Short Form will be used to retrospectively allocate participants to groups, with participants scoring ≥ + 1 standard error of the median on the Self-compassion Scale - Short Form allocated to a 'High self-compassion' group.
- 'Low self-compassion' group: Participants' total mean score on the Self-compassion Scale - Short Form (Raes et al., 2011) will be used as the independent variable. A median split (+/-1 standard error of the median) on the Self-compassion Scale - Short Form will be used to retrospectively allocate participants to groups, with participants scoring ≤ - 1 standard error of the median on the Self-compassion Scale - Short Form allocated to a 'Low self-compassion' group.

SUMMARY:
This study aims to investigate whether self-compassion is associated with older adult's quality of life after a diagnosis of dementia, and whether perceived threat posed by dementia mediates this relationship. Self-compassion has been found to be positive in supporting individuals in times of difficulty, in adjustment processes and older adults' wellbeing. While different factors have begun to be identified which are associated with individuals' psychological wellbeing and adjustment following a dementia diagnosis, little is known about the influence of self-compassion.

Participants will be recruited via NHS memory clinics, Join Dementia Research and from the community via third-sector organisations. Individuals will be invited to attend a Microsoft Teams/telephone appointment in which informed consent and cognitive screening processes will take place at the start. Eligible participants will then be invited to continue to complete measures administered by a researcher and an interview question. Participants will be offered the opportunity to complete the measures in a second session (within 8 weeks) or using the online survey software, Qualtrics, if preferred.

A small pilot study (n = 5) will take place prior to the main study.

ELIGIBILITY:
Inclusion Criteria:

* An older adult aged ≥ 65 years
* A confirmed diagnosis of dementia received within the past 12 months
* They have knowledge of their diagnosis
* They have English language proficiency
* They have capacity to give informed consent to participation.

Exclusion Criteria:

* They are deemed to lack capacity to give informed consent to participate (as per the Mental Capacity Act, 2005).
* They have a diagnosis of early-onset dementia, defined as individuals who are aged < 65 at diagnosis
* A score on the MoCA Blind (Nasreddine, 2022b) screening measure of <7 out of 22, which is calculated as equivalent to <10 out of 30 on the MoCA (Nasreddine et al., 2005).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The participant sample is anticipated to comprise NHS patients who have been seen in memory clinic and individuals recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Alzheimer's Disease (Logsdon et al., 1999) | Through study completion, average 40-60 minutes
  The Quality of Life in Alzheimer's Disease (Logsdon et al., 1999) consists of 13 items relating to different aspects of quality of life, such as mood, physical health, friends and ability to do things for fun. Each item is scored from 1 ('poor') to 4 ('excellent') to calculate a total score (Logsdon et al., 1999).

SECONDARY OUTCOMES:
Stress Appraisal Measure (Peacock and Wong, 1990) | Through study completion, average 40-60 minutes
  The Stress Appraisal Measure (Peacock & Wong, 1990) consists of 28 items pertaining to perceived future threat, measured across seven subscales; three referring to primary appraisals of threat, centrality and challenge, three relating to secondary appraisal - controllable by self, controllable by others and uncontrollable), and stressfulness. Only the threat and 'stressfulness' subscales, consisting of four items respectively, will be completed.
Geriatric Depression Scale - 10 (van Marwijk et al., 1995) | Through study completion, average 40-60 minutes
  The Geriatric Depression Scale - 10 (Van Marwijk et al., 1995), consisting of 10 items relating to how the person has felt over the past week (e.g. 'do you feel happy most of the time?'), has good reliability (α = 0.75), sensitivity and specificity (Almeida & Almeida, 1999). The Geriatric Depression Scale -10 is considered a reliable screening measure for major depression in older adults (Almeida & Almeida, 1999).

OTHER OUTCOMES:
Self-compassion Scale - Short Form (Raes, et al., 2011) | Through study completion, average 40-60 minutes
  The Self-Compassion Scale - Short Form (Self-Compassion Scale - Short Form; Raes et al., 2011) consists of 12 items relating to six subscales (self-judgement, self-kindness, common humanity, mindfulness, isolation and over-identification), with each item scored from 1 ('almost never') to 5 ('almost always') and three items reverse-scored. The Self-Compassion Scale - Short Form is a shortened version of the Self-Compassion Scale (Neff, 2003). Neff (2022) recommends utilising a total mean score calculated using the subscale mean scores, and this will be adopted in the current study to form the independent variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Health NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom